CLINICAL TRIAL: NCT01354262
Title: Does Vitamin D Supplement Alter Serum Level of Glycosylated Hemoglobin in Adult Patients Between 34-74 Years With Type 2 Diabetes Mellitus and Vitamin D Deficiency?
Brief Title: Effect of Vitamin D Supplementation on Hemoglobin A1c
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Prabhat Pokhrel, Physician, Ascension Health
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRMC 10 0023
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus; Vitamin D Deficiency
Keywords: Diabetes; Vitamin D deficiency; Hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lower dose vitamin D (Experimental): Fixed daily doses of 600 IU vitamin D oral supplementation.
  Interventions: Dietary Supplement: Vitamin D
- Higher dose vitamin D (Experimental): 50,000 IU supplementation bi-monthly.
  Interventions: Dietary Supplement: Vitamin D
- Control Group (No Intervention): Patients will be followed from baseline to 12 and 24 week follow up. Patients do not receive any research treatment or intervention beyond the standard care of their diabetes. This group are patients with normal levels of Vitamin D.

INTERVENTIONS:
Dietary Supplement: Vitamin D — 600 IU daily oral supplementation
  Arms: Lower dose vitamin D
Dietary Supplement: Vitamin D — 50,000 IU supplementation bi-monthly
  Arms: Higher dose vitamin D

SUMMARY:
This is a prospective, randomized, non-blinded interventional study that will investigate the effect of a vitamin D supplement on HbA1c in patients with uncontrolled type 2 diabetes mellitus (DM) and vitamin D deficiency. The goal is to investigate whether correcting vitamin D deficiency will alter the HbA1c level in patients with type 2 DM and lower than normal vitamin D level. My hypothesis is that correcting vitamin D deficiency decreases HbA1c levels in patients with type 2 DM and vitamin D deficiency.

DETAILED DESCRIPTION:
The total number of study subjects expected to be enrolled in this study is about 150. Study subjects included in this study will be men and women between 34-69 years of age who have been diagnosed with type 2 DM based on at least one of the American Diabetic Association criteria. These criteria are 1) fasting blood glucose higher than 125 mg/dL once with symptoms of diabetes (increased urination, increased appetite, increased thirst) or two times without symptoms; 2) random blood glucose more than 200 mg/dL once with symptoms or two times without symptoms of diabetes; 3) two hour glucose tolerance test more than 200 mg/dL once with symptoms or two times without symptoms; or 4) a random glycosylated hemoglobin more than 6.5 % two times. The age group for this research was selected based on the review of the literature on diabetes and vitamin D. Patients with known primary hyperparathyroidism, sarcoidosis, tuberculosis, cancer, potential terminal illness, history of serum creatinine more than 2.0 mg/dL, vitamin D supplement more than 200 IU/day, inflammatory bowel disease and history of hypercalcemia and kidney stones will be excluded from this study. For this project, vitamin D deficiency is defined as serum vitamin D level lower than 30 ng/mL and uncontrolled diabetes is defined as HbA1C level above 7.0. Although there is more than one recommended normal level of vit. D in the blood, most experts agree that the optimum serum level of vitamin D should be above 30 ng/mL. All subjects will be receiving standard of care for DM offered to them by his or her physician.

The investigators will investigate if different but fixed doses of vitamin D (600 IU a day vs 50,000 IU once every other week) when given to patients with type 2 DM and vitamin D deficiency have different effects on HbA1c level at the end of 24 weeks. A baseline blood draw, and fasting blood draws will be taken at 12 and 24 weeks for blood sugar levels, Vit D levels, and HgbA1c. Subjects with vitamin D deficiency will be randomly assigned to either group 1 or 2 and will be supplemented with either 600 IU of vitamin D/day (Group 1) or 50,000 IU of vitamin D every 2 weeks for 24 weeks (Groups 2). Patients who are not vitamin D deficient will be followed as the control group (Group 3) and will not be given any vitamin D supplement.Research subjects will be advised not to take any vitamin D or multivitamin while participating in this study. Subjects will be given 100 tablets of 600 IU of vitamin D in a bottle if they belong to Group 1. If they have been advised to take vitamin D 50,000 IU once every 14 days (Group 2), they will be given altogether 13 tablets of 50,000 of vitamin D each in a separate brown envelope with date written on the envelop and subjects will be asked to take vitamin D only on the date written on the envelop.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Hgb A1c greater then 7.0
* Adults aged 34 to 69 years.

Exclusion Criteria:

* known primary hyperparathyroidism, sarcoidosis, tuberculosis, cancer, potential terminal illness,
* history of serum creatinine more than 2.0 mg/dL,
* vitamin D supplement more than 200 IU/day
* history of inflammatory bowel disease, hypercalcemia or kidney stones

Ages: 34 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in serum levels of Hemoglobin A1c. | Change from baseline assessed at 12 wk and 24 wk.
  Serum levels of hemoglobin A1c will be tested in the laboratory from blood draws conducted at baseline and at 12 and 24 weeks from a fasting blood sample.

CONTACTS AND LOCATIONS:
Overall Officials: Prabhat K Pokhrel, MD, Principal Investigator — Ascension Health; Kimberly R Barber, PhD, Study Director — Ascension Health
Locations (1):
- Genesys East Flint Campus Clinic, Flint, Michigan, United States

REFERENCES:
- [Background] Avenell A, Cook JA, MacLennan GS, McPherson GC; RECORD trial group. Vitamin D supplementation and type 2 diabetes: a substudy of a randomised placebo-controlled trial in older people (RECORD trial, ISRCTN 51647438). Age Ageing. 2009 Sep;38(5):606-9. doi: 10.1093/ageing/afp109. Epub 2009 Jul 18. No abstract available. PMID 19617604
- [Background] Aljabri KS, Bokhari SA, Khan MJ. Glycemic changes after vitamin D supplementation in patients with type 1 diabetes mellitus and vitamin D deficiency. Ann Saudi Med. 2010 Nov-Dec;30(6):454-8. doi: 10.4103/0256-4947.72265. PMID 21060157